CLINICAL TRIAL: NCT04775277
Title: Outcome of Idiopathic Pulmonary Fibrosis With Pregnancy
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hend Mohammed Abdelraheem Esmaeel, assistant professor, Sohag University
Other Study IDs: Soh-Med-21-02-38
Record Dates: First submitted 2021-02-22; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: IPF; pregnancy
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: pregnant female with idiopathic pulmonary fibrosis
- control group: pregnant female with bronchial asthma

SUMMARY:
case-control study was conducted between December 2018 to April 2020. To document outcome of IPF with pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary diseases during pregnancy

Exclusion Criteria:

* Patients with pulmonary diseases other than IPF and bronchial asthma were excluded.

Ages: 18 Years to 38 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Female patients were diagnosed to have IPF of childbearing age, patients were presented during pregnancy
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
any adverse events including gestational complication or disease specific complication | from the start of inclusion to the study till termination of pregnancy, average 9 months period
  e.g (development of respiratory failure, need for ICU admission). maternal outcome
neonatal outcome | December 2018 to April 2020
  any unfavorable neonatal outcome as low birth weight
neonatal outcome | December 2018 to April 2020
  any unfavorable neonatal outcome as prematurity or neonatal death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Sharma CP, Aggarwal AN, Vashisht K, Jindal SK. Successful outcome of pregnancy in idiopathic pulmonary fibrosis. J Assoc Physicians India. 2002 Nov;50:1446-8. PMID 12583483